CLINICAL TRIAL: NCT04014049
Title: Assessment of the Relevance of a Medico-social Care of Elderly Patients, in Relay Between Hospital and Home: Experimentation of TEMPORARY HERBERGEMENT in Retirement Home " EHPAD " in Seine-et-Marne Department
Acronym: HT77
Status: Terminated | Type: Observational
Why Stopped: This study had to halt due to covid 19 pandemy.In fact, during the pandemy the two instutitions whose were included in this study were no longer accessible so this trial couldn't resume.In addition, the main criteria was invalidated by the pandemy.
Sponsor: Gérond'if (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A01189-48
Record Dates: First submitted 2019-07-07; First posted 2019-07-10 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Patients Beneficiting of Temporary Hebergement
Keywords: Temporary Hebergement (TH); Retirement Home (EHPAD); Discharge at home

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main objective is to study the impact of Temporary Hebergement (TH), as a medico-social care link between hospital and home, on the length of hospitalization in the referral services.

DETAILED DESCRIPTION:
It's a non-interventional, multi-centre study.

The request for Temporary Hebergement must be made by the principal investigator or on the recommendation of the other doctors in the co-investigator department at least 48 hours before the discharge from hospital. The EHPAD (Retirement Home) coordinating physician and/or nurse coordinator and the social worker plan the hospitalization release for Temporary Accommodation admission. The social worker must validate with the doctors the feasibility and coherence of the project of return to home, and write a summary attached to the admission file (social report) which will be used in the final analysis of the patients' return-to-home projects included in the study.

The hospital discharge for admission to HT is made with the agreement of the hospital doctor and the host EHPAD (Retirement home). A "check-list" is established to complete the patient's chart.

Upon admission and management of the patient in Temporary Hebergement , he will be followed by his treating physician. If necessary, the on-call doctor of the department that referred the patient may be contacted in case of hospital-applicant care. A mid-term review will be planned by the EHPAD (Retirement home social) worker to anticipate situations at risk of exit blockage at Day 30. The patient will be able to benefit from physiotherapy and speech therapy on prescription by liberal professionals working in the EHPAD, as well as occupational therapy and psychomotricity on the prescription of the coordinating physician during the development of the accompanying project. In addition, the Temporary Hebergement beneficiary will be able to participate in all the social activities of the residence, according to his wishes.

The following data: Quality of Life Questionnaire for Patients (Nottingham Scale) and Caregivers (SF-36 Scale), Caregiver Helper Questionnaire for Home Patients, Caregiver Burden Scale (Zarit) , ADL and IADL scales, EHPAD Patient and Caregiver Perception Questionnaire, Study Acceptability Questionnaire for Included Topics, Patient Comorbidity Evaluation Scale (Charlson) and Socio-Dataeconomic) are collected retrospectively, at Day 0 (inclusion), at Day 15, Day 30, Day 90 and Day 180 which corresponds to the end of the follow-up of patients provided for in the protocol

ELIGIBILITY:
Inclusion Criteria:

* Patient verbally expressing his non-opposition to participation in the study and documented in the medical record by the physician
* Hospitalized in hospitals selected as recruiting centers
* Whose condition is considered compatible by the clinician with discharge from the hospital (stabilized clinical condition)
* Resident, before hospitalization, in the department of Seine-et-Marne
* Presenting a defined and feasible return home project
* whose social situation does not allow an immediate return to the home on discharge from hospital

Exclusion Criteria:

* Patient expressing his opposition to participation in the study
* Acute condition not stabilized as per physician's medical opinion
* Requiring non-insured care by the host EHPAD, namely intravenous infusions, peritoneal dialysis, palliative care, etc.
* MMS score below 18
* Exhibiting behavioural disorders with major aggression and walking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving funded beds for "temporary accommodation" within EHPAD (Retirement Hom) recruiters.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
The main criterion used is the average length of stay (DMS) found at the end of the study, compared to the MSD for the two previous years in the services addressed. | 180 days

SECONDARY OUTCOMES:
Assessment of commorbidity risk according Charlson score | Inclusion , 2days
Assessment of teh degree of autonomy according AGGIR score | 180 days
Assessment of quality of life according "Nottingham health profile" scale | 180 days
Assessment of health-related quality of life according SF-36 (Medical outcome study Short-Form health survey-36 items) | 180 days
Assessment of the emotional, physical and financial burden on a caregiver according Zarit burden scale | 180 days
Assessment of the degree of patient dependence according "Index of Independence in Activities of Daily Living" KATZ scale | 180 days
Assessment of patient's level of dependence through an appreciation of instrumental activities of daily living according Lawton scale | 180 days

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Hanon, MD PhD, Study Chair — Geriatric Departement, Broca hospital, Paris
Locations (1):
- Geriatric department , Broca Hospital, Paris, Île-de-France Region, France